CLINICAL TRIAL: NCT00803881
Title: Prevalence of Chronic Rhinosinusitis, Pathogen-colonization in the Upper and Lower Airways and Ability to Smell in Cystic Fibrosis
Brief Title: Longitudinal Pathogen-colonization in Cystic Fibrosis Airways and Ability to Smell
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, PD Dr. Jochen G. Mainz, Head of CF Center, Pediatric Pulmonology, University of Jena
Other Study IDs: CF_Sinusitis_LS
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Cystic Fibrosis With Other Manifestations; Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Nasal Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CF patients of all age groups: Longitudinal prospective assessment of upper and lower airway colonization in all patients attended in the Jena University CF centre
  Interventions: Other: nasal lavage and sputum collection

INTERVENTIONS:
Other: nasal lavage and sputum collection — non-invasive longitudinal assessment of pathogen colonization in both airway levels
  Other Names: Pseudomonas aeruginosa antibodies in serum

SUMMARY:
Aim of the study is to detect the prevalence of chronic rhinosinusitis, pathogen colonization of the lower and upper airways and, in a sub-cohort the sense of smelling in patients with cystic fibrosis.

DETAILED DESCRIPTION:
The sub-study on the sense of smelling in CF has been finalized in the meantime. Results were published in 2012:

Smell in cystic fibrosis. Lindig J, Steger C, Beiersdorf N, Michl R, Beck JF, Hummel T, Mainz JG. Eur Arch Otorhinolaryngol. 2013 Mar;270(3):915-21. doi: 10.1007/s00405-012-2124-2. Epub 2012 Aug 14.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of cystic fibrosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients of the CF outpatients clinic and hospitalized CF patients
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2008-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Dynamics in CF upper and lower airway colonization with pathogens | 10 years
  longitudinal non-invasive sampling of upper and lower airways in CF
Assessment of ability to smell in CF patients | 3 years

SECONDARY OUTCOMES:
pulmonary function / BMI | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Mainz, MD, Study Chair — University of Jena - CF Center
Locations (1):
- University of Jena - CF-Center, Jena, Germany

REFERENCES:
- [Background] Lindig J, Steger C, Beiersdorf N, Michl R, Beck JF, Hummel T, Mainz JG. Smell in cystic fibrosis. Eur Arch Otorhinolaryngol. 2013 Mar;270(3):915-21. doi: 10.1007/s00405-012-2124-2. Epub 2012 Aug 14. PMID 22890694
- [Background] Mainz JG, Michl R, Pfister W, Beck JF. Cystic fibrosis upper airways primary colonization with Pseudomonas aeruginosa: eradicated by sinonasal antibiotic inhalation. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1089-90. doi: 10.1164/ajrccm.184.9.1089. No abstract available. PMID 22045752
- [Background] Mainz JG, Hentschel J, Schien C, Cramer N, Pfister W, Beck JF, Tummler B. Sinonasal persistence of Pseudomonas aeruginosa after lung transplantation. J Cyst Fibros. 2012 Mar;11(2):158-61. doi: 10.1016/j.jcf.2011.10.009. Epub 2011 Nov 30. PMID 22133899
- [Background] Mainz JG, Naehrlich L, Schien M, Kading M, Schiller I, Mayr S, Schneider G, Wiedemann B, Wiehlmann L, Cramer N, Pfister W, Kahl BC, Beck JF, Tummler B. Concordant genotype of upper and lower airways P aeruginosa and S aureus isolates in cystic fibrosis. Thorax. 2009 Jun;64(6):535-40. doi: 10.1136/thx.2008.104711. Epub 2009 Mar 11. PMID 19282318